CLINICAL TRIAL: NCT05212922
Title: An Open-Label, Non-Randomized, Multi-center Phase 2 Study of YH001 in Combination With Toripalimab in Subjects With Advanced Non-small Cell Lung Cancer (NSCLC) and Hepatocellular Carcinoma (HCC)
Brief Title: A Study to Evaluate YH001 in Combination With Toripalimab in Subjects With Advanced NSCLC and HCC
Acronym: YH001
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH001004
Record Dates: First submitted 2021-11-30; First posted 2022-01-28 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-11

CONDITIONS: HCC; NSCLC Stage IIIB; NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Single Group Assignmen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- YH001 + Toripalimab (Experimental): This study will include two cohorts of up to 40 subjects each treated with RP2D dose of YH001 in combination with 240 mg Toripalimab to assess the antitumor activity and safety/tolerability.
  Interventions: Drug: YH001 + Toripalimab

INTERVENTIONS:
Drug: YH001 + Toripalimab — YH001 + Toripalimab

SUMMARY:
This is an Open-label, Non-Randomized, Multi-center Phase 2 study of YH001 in Combination with Toripalimab，The study is designed to determine the safety ，tolerability and antitumor activity of YH001 in combination with Toripalimab in subjects with advanced NSCLC and HCC.

DETAILED DESCRIPTION:
This study will include two cohorts of up to 40 subjects each treated with RP2D dose YH001 in combination with 240 mg Toripalimab to assess the antitumor activity and safety/tolerability.

According to Simon's two stage design, in the first stage, 9-10 subjects will be accrued. If there are ≤ 1 subjects achieving an objective response, the futility stop will be called. Enrollment will start for the second stage after Stage 1 data pass futility test. In the second stage, 17-19 subjects will be enrolled to have 27 subjects in total. If there are ≥ 5 subjects achieving an objective response, a stop could be called for meeting the primary objective.

In all cohorts, 4 mg/kg or other higher dose level of YH001 (not exceeding MTD) may be needed based on the safety data in the first stage.

* Cohort A: YH001 in combination with Toripalimab in subjects with advanced PD-L1 positive NSCLC as 1st line treatment;
* Cohort B: YH001 in combination with Toripalimab in subjects with previously systemically treated advanced HCC as 2nd line treatment;

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years；
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Target Population

   Cohort A:
   * Have histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous)
   * Recurrent or unresectable locally advanced (Stage IIIB) or metastatic (Stage IV);
   * Naïve to any systemic anti-cancer therapy
   * No EGFR mutation or ALK/ ROS1 gene rearrangement
   * PD-L1 positive (TPS≥1%) NSCLC

   Cohort B:
   * HCC diagnosis confirmed by or radiology, histology, or cytology;
   * Barcelona Clinic Liver Cancer (BCLC) Stage C or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy and not amenable to a curative treatment approach;
   * Child-Pugh A liver score within 7 days prior to first dose of study drug;
   * Documented objective radiographic progression during or after treatment with sorafenib/lenvatinib, or intolerant of sorafenib/lenvatinib; or documented objective radiographic progression during or after treatment with atezolizumab and bevacizumab, or intolerant of atezolizumab and bevacizumab.
4. At least 1 unidimensional measurable target lesion per RECIST v1.1
5. ECOG performance status score 0 or 1
6. Have life expectancy of at least 12 weeks based on investigator's judgement.
7. Adequate organ and bone marrow function:
8. Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test within 7 days of the fist dose of YH001.
9. Women of reproductive potential who are sexually active with a non-sterilized male must consistently use highly effective contraception/birth control between signing of the informed consent and 120 days after the last administration of the study drug.

Exclusion Criteria:

1. Treatment with any investigational drug within 4 weeks prior to the fist dose of study drug；
2. Prior anticancer therapy:

   * Cohort B: Subjects received sorafenib/lenvatinib within 14 days of first dose of study medication.
   * Prior palliative radiotherapy to bone metastases ≤ 2 weeks prior to the first dose of YH001 is acceptable.
   * It is unacceptable to have wash out less than 2 weeks for herbal therapy approved for anticancer.
3. Subjects with prior anti-CTLA-4 checkpoint inhibitors should be excluded.
4. Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy or an AE of any grade that resulted in discontinuation of prior immunotherapy
5. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease
6. Subjects requiring systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 21 days before the planned first dose of study drug or has need to be treated while on trial
7. Allergic to YH001 and Toripalimab or any component of the study drug formulation.
8. Subjects with concomitant active autoimmune disease, history of autoimmune disease requiring systemic treatment, or history of autoimmune disease within the two years prior to study entry.
9. Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.
10. Subjects with severe cardiovascular diseases, e.g. New York Heart Association (NYHA) Class III or IV heart failure, myocardial infection within 6 months prior to first dose of YH001, uncontrolled hypertension, unstable angina pectoris or unstable cardiac arrhythmia.
11. QTcF > 470 ms at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome.
12. Viral infection:

    * Acute or Chronic active Hepatitis B (HBsAg positive and HBV DNA≥2000 IU/mL).
    * Chronic HCV infection (HCV antibody positive and HCV RNA detectable).
    * Human immunodeficiency virus (HIV) infection as well as COVID-19.
13. Subjects with active tuberculosis are excluded. Subjects who have received BCG vaccination may have a false positive PPD test. These subjects are eligible if they have a negative Interferon Gamma Release Assay (IGRA).
14. Clinically uncontrolled concurrent illnesses, including, but not limited to, active infection that requires systematic treatment, serious diabetes (fasting blood glucose > 250 mg/dl), psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies.
15. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that have not recovered to ≤ Grade 1 per CTCAE v5.0
16. Failure to recover adequately, as judged by the investigator, from prior surgical procedures; the subjects have had major surgery within 28 days, or minor surgery within 2 weeks prior to the first dose of YH001.
17. Subjects received any live or attenuated vaccine within 28 days prior to the first dosing of study drug. For inactivated or attenuated COVID -19 vaccine, follow local guidelines.
18. Pregnant or breast-feeding females.
19. Any clinically significant abnormality in the laboratory
20. Subjects have another active invasive malignancy within 5 years
21. Cohort B:

    * History of esophageal or gastric variceal bleeding within the last 6 months, or current active gastrointestinal bleeding;
    * Large tumor lesion in liver (≥60% liver volum), portal vein invasion at the main portal branch (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging;
    * Clinically diagnosed hepatic encephalopathy in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
ORR | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  Overall Response Rate (ORR) by investigator's assessment according to the RECIST v1.1

SECONDARY OUTCOMES:
safety and tolerability | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  The safety and tolerability will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
OS | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To assess other antitumor activity of YH001 in combination with Toripalimab
anti-drug antibodies (ADA) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  Immunogenicity
neutralizing antibodies (NAbs). | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To assess the immunogenicity of YH001 in combination with Toripalimab
peak concentration (Cmax) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To characterize the pharmacokinetic (PK) profiles of YH001 in combination with Toripalimab

OTHER OUTCOMES:
trough concentration (Ctrough) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To characterize the pharmacokinetic (PK) profiles of YH001 in combination with Toripalimab
terminal half-life (T1/2). | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To characterize the pharmacokinetic (PK) profiles of YH001 in combination with Toripalimab
Duration of response (DOR) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To assess other antitumor activity of YH001 in combination with Toripalimab by investigator's assessment according to the RECIST v1.1
progression free survival (PFS) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To assess other antitumor activity of YH001 in combination with Toripalimab by investigator's assessment according to the RECIST v1.1
time to response (TTR) | maximum of 1 years after the first dose of YH001 and Toripalimab study treatment.
  To assess other antitumor activity of YH001 in combination with Toripalimab by investigator's assessment according to the RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Rong Chen, Ph.D, Study Chair — Eucure (Beijing) Biopharma Co., Ltd
Locations (22):
- Gabrail Cancer Center Research, Canton, Ohio, Armenia
- Australia (2):
  - University of New South Wales (UNSW) - Liverpool Hospital, Liverpool, New South Wales
  - Andrew Love Cancer Centre, Geelong, Victoria
- Coffs Harbour Health Campus, Coffs Harbour, New South Wales, Austria
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The Affiliated Tumour Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Bethune First Hospital Of Jilin University, Changchun, Jilin
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
- Taiwan (7):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center - YongKang, Tainan
  - Chi Mei Medical Center - Liouying, Tainan
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No